CLINICAL TRIAL: NCT01407198
Title: Phase I Study of Nilotinib Given With Radiation For Patients With High Risk Chordoma
Brief Title: Nilotinib With Radiation for High Risk Chordoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Edwin Choy, MD, Instructor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-072
Record Dates: First submitted 2011-07-28; First posted 2011-08-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chordoma
Keywords: High Risk Chordoma
MeSH Terms: conditions — Chordoma | interventions — nilotinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib/XRT (Experimental): Nilotinib is administered 400mg PO BID for 2 weeks and then administered concurrently with daily radiation therapy until completion of radiation therapy. Participants can then undergo surgery if clinically possible. After either surgery or definitive radiation, participants have the option to continue on nilotinib therapy.
  Interventions: Drug: Nilotinib; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Nilotinib — Orally, daily 200 - 400 mg BID
  Other Names: AMN 107; Tasigna
Radiation: Radiation therapy — External beam radiation will be delivered at 1.8 Gy per day, 5 days per week (excluding holidays)for a total of 28 fractions over a 6 weeks period.
  Other Names: External beam radiation

SUMMARY:
The study drug, Nilotinib, is believed to slow down tumor growth by regulating a gene involved in cellular growth of chordoma cells. During this research study, subjects will also receive radiation therapy which is considered a standard treatment for advanced chordomas. It is hoped by adding nilotinib, the benefits of radiation therapy can be enhanced without adding significant toxicities.

The purpose of this research study is to determine the safety of nilotinib when used in combination with radiation therapy, and the highest dose of nilotinib that can be given safely with radiation therapy.

DETAILED DESCRIPTION:
Nilotinib will be taken orally daily in two cycles of 28 days each. Two weeks after taking nilotinib, subjects will begin radiation therapy. Radiation therapy will continue every weekday until Day 56 of the study. If it is determined that the subject's tumor cannot be removed by surgery, an additional 3 weeks of radiation therapy will be applied after Day 56 of the study.

During study visits subjects will have physical exams, routine blood tests, urine and blood clotting tests, and EKGs. Subjects will also have tumor assessment by chest CT and MRI or CT of the tumor at screening, on approximately Day 56 of the study, then every 6 months for one year and then annually thereafter if ther is no disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chordoma
* Considered to have high risk disease
* Measurable disease
* Life expectancy > 3 months
* Adequate organ function
* Able to swallow oral capsules

Exclusion Criteria:

* Previous treatment with any other tyrosine kinase inhibitor
* Previous treatment with radiotherapy to the primary or recurrent chordomas
* Impaired cardiac function
* Currently receiving treatment with strong CYP3A4 inhibitors
* Requires anticoagulation with coumadin
* Impaired GI function or GI disease that may significantly alter the absorption of study drug
* Acute or chronic pancreatic disease
* Known cytopathologically confirmed CNS infiltration
* Another primary malignant disease which requires systemic treatment
* Acute or chronic liver disease or severe renal disease considered unrelated to the cancer
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Major surgery within 4 weeks prior to Day 1 of the study or who have not recovered from prior surgery
* Treatment with other investigational agents within 30 days of Day 1
* History of non-compliance to medical regimens
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2016-02 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities (DLTs) for participants when treated above the maximum tolerated dose (MTD). | 2 years
  A DLT will be defined as any of the following events occurring during days 1-56 of study according to CTCAE version 4.0. MTD is then determined by identifying a dose cohort demonstrating > or = 30% rate of DLTs, which are defined as:
  * Any Grade ≥ 3 nonhematologic toxicity except alopecia, nausea, or vomiting not otherwise controlled by maximual supportive care.
  * Grade 4 neutropenia (ANC < 500/µL) lasting > 5 days, Grade 3 thrombocytopenia lasting > 7 days, or Grade 4 thrombocytopenia
  * Failure to resume treatment delays within a defined period of time.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 2 years
  Adverse event profile, as determined by CTC AE version 4.0, will be determined for patients treated with nilotinib and radiation therapy.
  Adverse events analyses will include:
  * Detailed examination of adverse events
  * Laboratory test results
  * Vital signs or other physical findings
  * Frequency and extent of dose modification
  The assessment of adverse events will be based mainly on the frequency of adverse events, particularly adverse events leading to discontinuation of treatment and on the number of significant laboratory abnormalities.
Survival | 2 years
  To obtain preliminary data regarding local control, distant control, disease-free survival, and overall survival with this regimen
PDGFR signaling | 2 years
  To determine if nilotinib decreases PDGFR signaling in chordoma tumor samples in treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Choy, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No